CLINICAL TRIAL: NCT03936036
Title: Replication of the CARMELINA Diabetes Trial in Healthcare Claims
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-CARMELINA
Record Dates: First submitted 2019-04-29; First posted 2019-05-03 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Linagliptin; Sulfonylurea Compounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2nd generation sulfonylureas: Reference group
  Interventions: Drug: Sulfonylurea
- Linagliptin: Exposure group
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: Linagliptin — Linagliptin dispensing claim is used as the exposure
  Groups: Linagliptin
Drug: Sulfonylurea — 2nd generation sulfonylurea dispensing claim is used as the reference
  Groups: 2nd generation sulfonylureas

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see: https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Eligible cohort entry dates Market availability of linagliptin in the U.S. started on May 2, 2011. For Marketscan and Medicare: May 2, 2011-Dec 31, 2016 (end of data availability).

For Optum: May 2, 2011-Sep 30, 2017 (end of data availability).

Inclusion Criteria:

1. Documented diagnosis of T2DM before visit 1 (screening).
2. Male or female patients who are drug-naïve or pre-treated with any antidiabetic background therapy, excluding treatment with GLP-1 receptor agonists, DPP-4 inhibitors or SGLT-2 inhibitors if ≥ 7 consecutive days.
3. Stable antidiabetic background medication (unchanged daily dose) for at least 8 weeks prior to randomization. If insulin is part of the background therapy, the average daily insulin dose should not have been changed by more than 10% within the 8 weeks prior to randomization compared with the daily insulin dose at randomization.
4. HbA1c of ≥ 6.5% and ≤ 10.0% at visit 1 (screening).
5. Age ≥ 18 years at visit 1 (screening). For Japan only: Age ≥ 20 years at Visit 1.
6. Body Mass Index (BMI) 45 kg/m2 at visit 1 (screening).
7. Signed and dated written informed consent by date of visit 1 (screening) in accordance with GCP and local legislation prior to any study related procedure.
8. High risk of CV events (I and/or II):

Albuminuria (UACR ≥ 30 mg/g creatinine or ≥ 30 µg/min [microgram albumin per minute] or ≥ 30 mg/24 h [milligram albumin per 24 hours] in two out of three unrelated spot urine or timed samples in the last 24 months prior to randomization)*

AND previous macrovascular disease, defined as either one or more:

Confirmed history of MI (> 2 months prior to Visit 1)

Advanced coronary artery disease, defined by any one of the following:

* ≥ 50% narrowing of the luminal diameter in 2 or more major coronary arteries by coronary angiography, MRI angiography or CT angiography; Definition of major coronary arteries: LAD (Left Anterior Descending). CX (Circumflex) or RCA (right coronary artery)
* Left main stem coronary artery with ≥ 50% narrowing of the luminal diameter by coronary angiography, MRI angiography or CT angiography;
* Prior percutaneous or surgical revascularization of 2 major coronary arteries at least 2 months prior to Visit 1 (screening);
* The combination of prior percutaneous or surgical revascularization of 1 major coronary artery at least 2 months prior to visit 1 (screening), and ≥ 50% narrowing of the luminal diameter by coronary angiography, MRI angiography or CT angiography of at least 1 additional major coronary artery.

  10) High-risk single-vessel coronary artery disease, defined as the presence of 50% narrowing of the luminal diameter of one major coronary artery by coronary angiography, MRI angiography or CT angiography in patients not revascularised:

AND at least one of the following:

* A positive non invasive stress test, confirmed by either:
* a positive ECG exercise tolerance test in patients without left bundle branch block, Wolff-Parkinson-White syndrome, left ventricular hypertrophy with repolarization abnormality, or paced ventricular rhythm, atrial fibrillation in case of abnormal ST-T segments;
* a positive stress echocardiogram showing induced regional systolic wall motion abnormalities;
* a positive nuclear myocardial perfusion imaging stress test showing stress- induced reversible perfusion abnormality;
* a positive cardiac stress perfusion MRI showing a stress induced perfusion defect;
* Patient discharged from hospital with a documented diagnosis of unstable angina pectoris between 2 and 12 months prior to visit 1 (screening).

  10) History of ischemic or haemorrhagic stroke (>3 months prior to visit 1) 11) Presence of carotid artery disease (symptomatic or not) documented by either:
* imaging techniques with at least one lesion estimated to be ≥50% narrowing of the luminal diameter;
* prior percutaneous or surgical carotid revascularization. 12) Presence of peripheral artery disease documented by either:
* previous limb angioplasty, stenting or bypass surgery;
* previous limb or foot amputation due to macrocirculatory insufficiency;
* angiographic evidence of peripheral artery stenosis 50% narrowing of the luminal diameter in at least one limb (definition of peripheral artery: common iliac artery, internal iliac artery, external iliac artery, femoral artery, popliteal artery).

  13) Evidence of impaired renal function with predefined UACR, with or without CV co- morbidities, defined as follows (and/or criteria):
  * Impaired renal function (as defined by MDRD formula) with an eGFR: 15- <45 mL/min/1.73 m2 at visit 1 (screening) with any UACR.
  * Impaired renal function (as defined by MDRD formula) with an eGFR ≥ 45-75 mL/min/1.73 m2 at visit 1 (screening) with an UACR > 200 mg/g creatinine or > 200 µg/min (microgram albumin per minute) or > 200 mg/24 h [milligram albumin per 24 hours] demonstrated in two out of three unrelated spot urine or timed samples in the last 24 months prior to randomization.

Exclusion Criteria:

1. Type 1 diabetes mellitus.
2. Treatment (≥ 7 consecutive days) with GLP-1 receptor agonists, other DPP-4 inhibitors or SGLT-2 inhibitors prior to informed consent. Note: This also includes clinical trials where these antidiabetic drugs have been provided to the patient.
3. Active liver disease or impaired hepatic function, defined by serum levels of either ALT (SGPT), AST (SGOT), or alkaline phosphatase (AP) ≥3 x upper limit of normal (ULN) as determined at Visit 1.
4. eGFR <15 ml/min/1.73 m2 (severe renal impairment or ESRD, MDRD formula), as determined during screening at Visit 1 and/or the need for maintenance dialysis.
5. Any previous (or planned within next 12 months) bariatric surgery (open or laparoscopic) or intervention (gastric sleeve).
6. Pre-planned coronary artery re-vascularisation (PCI, CABG) or any previous PCI and/or CABG ≤ 2 months prior informed consent"
7. Known hypersensitivity or allergy to the investigational products or its excipients.
8. Any previous or current alcohol or drug abuse that would interfere with trial participation in the opinion of the investigator.
9. Participation in another trial with an investigational drug ongoing or within 2 months prior to visit 1 (screening)*.
10. Pre-menopausal women (last menstruation 1 year prior to informed consent) who:

    * are nursing or pregnant,
    * or are of child-bearing potential and are not practicing an acceptable method of birth control (acceptable methods of birth control include tubal ligation, transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, sexual abstinence (if allowed by local authorities), double barrier method and vasectomised partner) or do not plan to continue using acceptable method of birth control throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial.
11. Patients considered unreliable by the investigator concerning the requirements for follow- up during the study and/or compliance with study drug administration, have a life expectancy less than 5 years for non-CV causes, or have cancer other than non-melanoma skin cancer within last 3 years, or has any other condition than mentioned which in the opinion of the investigator, would not allow safe participation in the study."
12. Acute coronary syndrome (ACS), diagnosed ≤ 2 months prior to visit 1 (screening).
13. Stroke or TIA ≤ 3 months prior to visit 1 (screening).

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, cohort study design comparing linagliptin to the 2nd generation sulfonylurea (SU) antidiabetic class as a proxy for placebo. SUs are not known to have an impact on the outcome of interest. In addition, SUs were the most frequent background treatment in CARMELINA (after metformin), and DPP4i and SUs are preferentially prescribed to similarly older patients in real world (Patorno et al., 2019). The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of linagliptin or a comparator drug (cohort entry date). Follow-up for the outcome (3P-MACE), begins the day after drug initiation. As in the trial, patients are allowed to take other antidiabetic medications during study follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 101830 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Relative hazard of composite outcome of Stroke, MI, and Mortality | Through study completion (a median of 118-123 days)
  Relative hazard of composite outcome of MI, stroke, and mortality - Please refer to uploaded protocol for full definition due to size limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Franklin JM, Patorno E, Desai RJ, Glynn RJ, Martin D, Quinto K, Pawar A, Bessette LG, Lee H, Garry EM, Gautam N, Schneeweiss S. Emulating Randomized Clinical Trials With Nonrandomized Real-World Evidence Studies: First Results From the RCT DUPLICATE Initiative. Circulation. 2021 Mar 9;143(10):1002-1013. doi: 10.1161/CIRCULATIONAHA.120.051718. Epub 2020 Dec 17. PMID 33327727

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT03936036/Prot_SAP_002.pdf